CLINICAL TRIAL: NCT01375296
Title: China Made Sirolimus Eluting Stent for Treatment of Coronary Intermediate Lesion
Brief Title: China Made Sirolimus Eluting Stent for Intermediate Lesion
Acronym: SESIL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Weifeng Shen, Ruijin hospital, shanghai jiao tong university school of medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJH20100918
Record Dates: First submitted 2011-04-01; First posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- SES (Experimental): including two types of China-made SES, i.e. Firebird 2 (cobalt-alloy platform with durable polymer coating sirolimus-eluting stent) and Excel (stainless steel platform with biodegradable polymer coating sirolimus-eluting stent).
  Interventions: Device: China-made SES (Firebird 2 and Excel)
- medicine (Other)
  Interventions: Other: routine medicine

INTERVENTIONS:
Device: China-made SES (Firebird 2 and Excel) — patients with coronary 50-70% narrowing treated with China-made SES stent,i.e. Firebird 2 (cobalt-alloy platform with durable polymer coating sirolimus-eluting stent) and Excel (stainless steel platform with biodegradable polymer coating sirolimus-eluting stent).
  Arms: SES
Other: routine medicine — patients with coronary 50-70% narrowing treated with routine medicine
  Arms: medicine

SUMMARY:
Sirolimus-eluting stent (SES) has been proven to improve outcomes in patients with significant coronary artery diseae(> 70% lumen diameter narrowing). But, acute coronary syndrome may occur in those with intermediate lesions(50%-70% lumen diameter narrowing), and the effect of SES in these patients remains unclear. Here the investigators hypothesize that application of China-made SES may improve the clinical outcomes in these setting.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old
* both gender
* native coronary lesion
* narrowing 50-70%
* vessel size 2.5-4.0 in diameter

Exclusion Criteria:

* without informed consent,
* ST elevation myocardial infarction within 7 days,
* left main lesion,
* by-pass graft,
* restenosis
* abnormal liver function before randomization,
* active hepatitis or muscular disease,
* impaired renal function with serum creatinine level > 3mg/dl ,
* impaired left ventricular function with LVEF < 30%,
* participate in other studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
target vessel failure | 12 months
  defined as the occurrence of any of the following within 12 months after the index procedure: death from cardiac causes, Q-wave or non-Q-wave myocardial infarction, or revascularization of the target vessel (emergency or elective coronaryartery bypass grafting [CABG] or repeated percutaneous transluminal coronary angioplasty [PTCA]).

SECONDARY OUTCOMES:
major adverse cardiac events | 12 months
  including cardiac death, re-infarction and target vessel revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- ruijin hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China